CLINICAL TRIAL: NCT01108315
Title: Phase II Study of Comprehensive Patient Reported Outcomes (PRO) Management for Oncology Practice
Brief Title: Comprehensive Patient Reported Outcomes (PRO) Management for Oncology Practice
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BrightOutcome (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Niina Haas, Project Director, BrightOutcome
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HC4ext; NCI (Other Grant/Funding Number: HHSN261200700046C)
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: Patient Reported Outcomes (PRO); Web-based; Phone-based; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The participant used the web and/or phone-based PRO reporting symptoms to enter symptoms twice a week at minimum.
  Interventions: Other: Report symptoms via web or phone-based system
- Usual Care (No Intervention): The participants on this arm do not record their symptoms. They report symptoms as they would under usual care.

INTERVENTIONS:
Other: Report symptoms via web or phone-based system — The participant reports their symptoms at least twice a week via the phone or web-based prototype system.
  Arms: Intervention

SUMMARY:
Cancer symptoms due to disease progression or side effects caused by cancer treatment are prevalent. Most cancer patients are treated in outpatient settings. Patients may be provided with patient education materials and counseled on anticipated side effects while being provided with different self-management options and warnings regarding when medical care is required. Despite these efforts, many people feel set adrift in having to self-manage treatment and illness related symptoms at home resulting in a sense of burden for the patient and the caregiver.

When the patient does visit the doctor, they increasingly are asked questions to elicit information about symptoms and performance using structured questionnaires that are shown to give reproducible, meaningful, quantitative assessments of how patients feel and how they function-measures that are called patient reported outcomes or PROs. The questionnaires used to collect this information are called PRO instruments. The use of PRO instruments is part of a general movement toward the idea that the patient, properly queried, is the best source of information about how he or she feels. The goal of using PRO measures is to provide better information to doctors and patients so that the best treatment for patients can be determined.

PURPOSE: To reduce the isolation of patients/caregivers from the medical care team and to improve patient/provider communication and clinical decisions by keeping documented daily reports of patient symptoms online, having notifications sent to the medical team of moderate to severe symptoms and by reviewing these reports at clinic visits with the medical staff.

ELIGIBILITY:
Inclusion Criteria:

* Female, breast oncology patient
* Breast cancer diagnosis
* Expected chemotherapy regimen of at least 3-4 months
* Sufficient cognitive ability and psychological stability in the opinion of treating physician
* Fluent in spoken and written English
* 18 years of age or older
* Outpatient
* Life expectancy > 6 months as estimated by treating physician
* Informed of the investigational nature of this study and provided informed consent.
* Has access to either a phone or the internet

Exclusion Criteria:

* Is not female, nor a breast oncology patient
* Does not have breast cancer diagnosis
* Expected chemotherapy regimen is less than 3-4 months
* Does not have sufficient cognitive ability and psychological stability in the opinion of treating physician
* Is not fluent in spoken and written English
* Is younger than 18 years of age
* Inpatient
* Life expectancy < 6 months as estimated by treating physician
* Is not informed of the investigational nature of this study and does not provide informed consent.
* Does not have access to either a phone or internet.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Usability and effectiveness of the prototype | 6 months
  Usability and effectiveness of BrightOutcome's web and phone-based symptom reporting and assessment software as it pertains to patient/provider communication

CONTACTS AND LOCATIONS:
Overall Officials: DerShung Yang, PhD, Principal Investigator — BrightOutcome; VK Gadi, MD, Principal Investigator — University of Washington; Ana Maria Lopez, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Arizona Cancer Center, Tucson, Arizona
  - Seattle Cancer Care Alliance, Seattle, Washington